CLINICAL TRIAL: NCT00329628
Title: RECORD 1 Study: REgulation of Coagulation in ORthopedic Surgery to Prevent DVT and PE, Controlled, Double-blind, Randomized Study of BAY 59-7939 in the Extended Prevention of VTE in Patients Undergoing Elective Total Hip Replacement
Brief Title: Rivaroxaban (10mg) Given Once Daily in Patients Undergoing Total Hip Replacement Compared to Enoxaparin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11354; EudraCT: 2005-004351-35
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Venous Thromboembolism
Keywords: Prevention; Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism; Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)
- Arm 2 (Active Comparator)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Rivaroxaban (BAY59-7939) — 10 mg OD tablet of rivaroxaban administered for 36 +/- 4 days
  Arms: Arm 1
Drug: Enoxaparin — Syringe of Enoxaparin active substance at a dose of 40 mg administered for 13 +/- 2 days
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess if 10 mg BAY 59-7939, taken once daily as a tablet, is safe and prevent blood clot which may form after total hip replacement operation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years or above
* Patients scheduled for elective total hip replacement

Exclusion Criteria:

* Planned, staged total bilateral hip replacement
* Active bleeding or high risk of bleeding contraindicating treatment with low molecular weight heparin
* Contraindication listed in the labeling or conditions precluding patient treatment with enoxaparin
* Conditions prohibiting bilateral venography (e.g. amputation of one leg, allergy to contrast media)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4541 (Actual)
Dates: Start 2006-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of total VTE i.e.: Any DVT (proximal and/or distal), Non fatal PE, Death of all causes | Treatment period : up to day 36+/-6

SECONDARY OUTCOMES:
Incidence of the composite endpoint comprising proximal DVT, non-fatal PE and VTE- related death (major VTE) | Treatment period : up to day 36+/-6
Incidence of symptomatic VTE (DVT, PE) | Treatment period : up to day 36+/-6
Incidence of DVT (total, proximal, distal) | Treatment period : up to day 36+/-6
Incidence of symptomatic VTE during follow-up | Follow-up period: following 36+/-6 days
The composite endpoint comprising major VTE and treatment-emergent major bleeding | For major VTE, treatment period: up to Day 36+/-6 ; for major bleeding, from first dose of double-blind study medication to up to two days after last dose of double-blind study medication
Incidence of the composite endpoint that results from the primary endpoint by substituting VTE related death for all death | Treatment period : up to day 36+/-6
Incidence of the composite endpoint that results from major VTE by substituting all cause mortality for VTE-related death | Treatment period : up to day 36+/-6
Treatment-emergent major bleedings | From first dose of double-blind study medication to up to two days after last dose of double-blind study medication

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (188):
- United States (13):
  - Birmingham, Alabama
  - Northport, Alabama
  - Phoenix, Arizona
  - Benton, Arkansas
  - La Jolla, California
  - Aurora, Colorado
  - Decatur, Georgia
  - Missoula, Montana
  - Charleston, South Carolina
  - Dallas, Texas
  - Grapevine, Texas
  - Lubbock, Texas
  - San Antonio, Texas
- Argentina (3):
  - Avellaneda, Buenos Aires
  - Berazategui, Buenos Aires
  - Buenos Aires, Buenos Aires F.D.
- Australia (4):
  - Sydney, New South Wales
  - Adelaide, South Australia
  - Melbourne, Victoria
  - Fremantle, Western Australia
- Austria (7):
  - Wiener Neustadt, Lower Austria
  - Graz, Styria
  - Innsbruck, Tyrol
  - Linz, Upper Austria
  - Ried, Upper Austria
  - Wels, Upper Austria
  - Vienna, Vienna
- Belgium (10):
  - Antwerp
  - Brasschaat
  - Bruges
  - Genk
  - Hasselt
  - Huy
  - Merksem
  - Pellenberg
  - Reet
  - Roeselare
- Brazil (3):
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Canada (8):
  - Edmonton, Alberta
  - Kitchener, Ontario
  - Oakville, Ontario
  - Oshawa, Ontario
  - Peterborough, Ontario
  - Stratford, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Santiago, Chile
- Bogotá, Colombia
- Czechia (10):
  - České Budějovice
  - Hradec Králové
  - Jindřichův Hradec
  - Karlovy Vary
  - Mladá Boleslav
  - Olomouc
  - Pilsen
  - Prague
  - Pribram I
  - Prostějov
- Denmark (5):
  - Frederiksberg
  - Hellerup
  - Herlev
  - Hørsholm
  - Silkeborg
- Finland (3):
  - Jyväskylä
  - Mikkeli
  - Seinäjoki
- France (10):
  - Bois-Guillaume
  - Le Chesnay
  - Liévin
  - Monaco
  - Nantes
  - Paris
  - Saint-Herblain
  - Soyaux
  - Vandœuvre-lès-Nancy
  - Vannes
- Germany (17):
  - Bad Mergentheim, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Rheinfelden, Baden-Wurttemberg
  - Stuttgart, Baden-Wurttemberg
  - Fürth, Bavaria
  - Garmisch-Partenkirchen, Bavaria
  - Würzburg, Bavaria
  - Birkenwerder, Brandenburg
  - Sommerfeld, Brandenburg
  - Bremen, City state Bremen
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Wiesbaden, Hesse
  - Rostock, Mecklenburg-Vorpommern
  - Düsseldorf, North Rhine-Westphalia
  - Witten, North Rhine-Westphalia
  - Dresden, Saxony
- Greece (2):
  - Haidari, Attica
  - Kifissia, Attica
- Hungary (8):
  - Kaposvár, Hungary
  - Békéscsaba
  - Budapest
  - Győr
  - Kecskemét
  - Szeged
  - Szekszárd
  - Székesfehérvár
- Israel (8):
  - Beersheba, Israel
  - Haifa, Israel
  - Holon, Israel
  - Kfar Saba, Israel
  - Petah Tikva, Israel
  - Tel Aviv, Israel
  - Ẕerifin, Israel
  - Tel Litwinsky
- Italy (19):
  - Monza, Milano
  - Rozzano, Milano
  - San Donato Milanese, Milano
  - Gubbio, Perugia
  - Alghero, Sassari
  - Busto Arsizio, Varese
  - Ancona
  - Bergamo
  - Bologna
  - Ferrara
  - Florence
  - Genova
  - Milan
  - Palermo
  - Reggio Emilia
  - Roma
  - Sassari
  - Torino
  - Varese
- Lithuania (2):
  - Kaunas
  - Vilnius
- Mexico (2):
  - Monterrey, Nuevo León
  - Edo. de Mexico
- Netherlands (7):
  - Amsterdam
  - Hilversum
  - Hoofddorp
  - Leiden
  - Nijmegen
  - Oss
  - Zwolle
- Norway (5):
  - Baerum Postterminal
  - Elverum
  - Gjøvik
  - Lillehammer
  - Notodden
- Poland (13):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Opole
  - Poznan
  - Sosnowiec
  - Szczecin
  - Warsaw
  - Wroclaw
- Slovakia (3):
  - Kosice - Saca, Slovakia
  - Bratislava
  - Žilina
- South Africa (3):
  - Pretoria, Gauteng
  - Somerset West, Western Cape
  - Worcester, Western Cape
- Spain (12):
  - Santiago de Compostela, A Coruña
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Castellon, Castellón de La Plana
  - Jaén, Jaén
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Pamplona, Pamplona
  - Oviedo, Principality of Asturias
  - Valencia, Valencia
  - Vitoria-Gasteiz, Vitoria
- Sweden (6):
  - Gothenburg
  - Halmstad
  - Jönköping
  - Lidköping
  - Varberg
  - Västervik
- Turkey (Türkiye) (3):
  - Adana
  - Istanbul
  - Izmir

REFERENCES:
- [Derived] Eriksson BI, Borris LC, Friedman RJ, Haas S, Huisman MV, Kakkar AK, Bandel TJ, Beckmann H, Muehlhofer E, Misselwitz F, Geerts W; RECORD1 Study Group. Rivaroxaban versus enoxaparin for thromboprophylaxis after hip arthroplasty. N Engl J Med. 2008 Jun 26;358(26):2765-75. doi: 10.1056/NEJMoa0800374. PMID 18579811
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu